CLINICAL TRIAL: NCT02583841
Title: "Effect of Scaling and Root Planing on Liver Function Test (Alanine Aminotransferase and Aspartate Aminotransferase) in Systemically Healthy - Chronic Periodontitis Subjects: a Clinical Trial."
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr. Pradnya Rajendra Khatavkar, Post graduate student, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TatyasahebKoreDentalC
Record Dates: First submitted 2015-10-17; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Periodontitis (CP) Subjects.
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Scaling and Root Planing( SRP) (Active Comparator): This was an interventional study in which scaling and root planing was done in systemically healthy patients with chronic periodontitis
  Interventions: Procedure: Scaling and root planing
- Control Group (No Intervention): Scaling and root planing was not done , that is no intervention is carried out in the patients of this group.

INTERVENTIONS:
Procedure: Scaling and root planing — scaling and root planing as an intervention was done in patients of the test group
  Arms: Scaling and Root Planing( SRP)

SUMMARY:
Aim:

To evaluate effect of non- surgical periodontal therapy on liver function in systemically healthy chronic periodontitis (CP) subjects.

Materials and methods:

The study is non surgical interventional trial, includes 50 CP subjects in the age group of 35- 60 years selected from the OPD (Out Patient Department) of department of periodontology Tatyasaheb Kore Dental College and Research center (TKDC and RC), Kolhapur. CP subjects were equally divided into test group and control group. Liver function test- aspartate aminotransferase (AST), alanine aminotransferase (ALT) were checked at baseline and at 1 month after treatment. Clinical examination includes plaque index, gingival index, sulcus bleeding index, probing depth, clinical attachment loss.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with CP (moderate and severe) as per Centers for disease control and prevention (CDC) criteria 2007.
2. Patients without any known systemic diseases

   -

Exclusion Criteria:

1. Patients who have taken anti-inflammatory/antibiotic/antioxidant within 3 months of beginning of study.
2. Subjects who have undergone periodontal treatment within six months of inception of study.
3. Smokers, tobacco habits in any form and alcoholics.
4. Pregnant and lactating women.

   -

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Alanine aminotransferase | 1month
Aspartate aminotransferase | 1 month

SECONDARY OUTCOMES:
plaque index | 1month
gingival index | 1 month
sulcus bleeding index | 1month
probing depth | 1month
Clinical attachment loss | 1 month